CLINICAL TRIAL: NCT07307482
Title: Study on the Mechanism of Gut Microbiota Mediating Restless Legs Syndrome Through Iron Metabolism
Status: Not yet recruiting | Type: Observational
Sponsor: Wenxia Jiang (Other)
Responsible Party: Sponsor-Investigator, Wenxia Jiang, Doctor, Chongqing Traditional Chinese Medicine Hospital
Organization: Chongqing Traditional Chinese Medicine Hospital (Other)
Other Study IDs: 2025-IIT-KS-23
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Restless Legs Syndrome (RLS)
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
The goal of this observational study is to collect fecal and serum samples from patients with restless legs syndrome (RLS) and healthy controls for differential microbiota analysis to identify key bacterial species involved in the pathogenesis of RLS. Subsequently, metabolomic analysis will be performed on fecal and serum samples from RLS patients to identify key regulatory molecules in iron metabolism disorder pathways. Finally, correlation analysis will be used to determine which specific bacterial species and metabolites are involved in the pathogenesis of RLS. The main question it aims to answer is: i) Do RLS patients exhibit gut microbiota dysbiosis compared to healthy controls? ii) Which specific bacterial species and metabolites are linked to iron metabolism abnormalities and the pathogenesis of RLS?

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* The diagnostic criteria all meet the five diagnostic criteria for restless legs syndrome established by the International Committee for the Study of Restless Legs Syndrome (IRLSSG) (2014 revised version)

Exclusion Criteria:

* Suffering from serious physical illnesses, such as tumors, cardiovascular diseases, diabetes, stroke, etc.;
* Drug abuse, alcoholism, acute poisoning;
* Antibiotic use within the 4 weeks preceding sampling;
* Arobiotics or prebiotics use within the 4 weeks preceding sampling;
* Iron supplements use within the 4 weeks preceding sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 50 patients with restless legs syndrome from among those attending the Sleep Medicine Center of Chongqing Traditional Chinese Medicine Hospital during the period December 2025 to December 2026.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
There are differences in the abundance of gut microbiota between RLS and theThere are differences in the abundance of gut microbiota between RLS patients and the healthy controls. | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Yan, F., Y. Cheng, and S. Feng, Association between serum GFAP, BDNF and NfL levels and clinical symptoms in restless legs syndrome: a case-control study. Sleep Med, 2025. 134: p. 106694. 2. Holland, M.T., et al., Adaptive spinal cord stimulation improves restless legs syndrome: Case report, literature review, and mechanistic hypothesis. Sleep Med, 2025. 134: p. 106664. 3. Takahara, I., et al., Prevalence of Restless Legs Syndrome in Patients with Inflammatory Bowel Disease. Dig Dis Sci, 2017. 62(3): p. 761-767. 4. Loosen, S.H., et al., Association between Inflammatory Bowel Disease and Subsequent Development of Restless Legs Syndrome and Parkinson's Disease: A Retrospective Cohort Study of 35,988 Primary Care Patients in Germany. Life (Basel), 2023. 13(4). 5. Hackethal, S., et al., Restless Legs Syndrome During Pregnancy and Puerperium. Sleep, 2025. 6. Elangovan, P., et al., Prevalence of Restless Leg Syndrome and Its Association With Iron Deficiency in Patients With Chronic Kidney Disease: A Cross-Sectional Observational Study. Cureus, 2025. 17(6): p. e86188. 7. Schormair, B., et al., Genome-wide meta-analyses of restless legs syndrome yield insights into genetic architecture, disease biology and risk prediction. Nat Genet, 2024. 56(6): p. 1090-1099. 8. Manconi, M., et al., Restless legs syndrome. Nat Rev Dis Primers, 2021. 7(1): p. 80. 9. Guo, X., et al., Clinical feature and alpha-synuclein level of restless legs syndrome with leucine-rich repeat kinase 2 encoding gene mutation. Parkinsonism Relat Disord, 2025. 138: p. 107944. 10. Earley, C.J., et al., Altered brain iron homeostasis and dopaminergic function in Restless Legs Syndrome (Willis-Ekbom Disease). Sleep Med, 2014. 15(11): p. 1288-301. 11. Mizuno, S., et al., CSF iron, ferritin and transferrin levels in restless legs syndrome. J Sleep Res, 2005. 14(1): p. 43-7. 12. Ferré, S., et al., New Insights into the Neurobiology of Restless Legs Syndrome. Neuroscientist, 2019. 25(2): p. 113-125.